CLINICAL TRIAL: NCT03153358
Title: Icotinib Combined With Stereotactic Body Radiation Therapy (SBRT) for Patients With Metastatic Non-squamous Non-small Cell Lung Cancer With EGFR Sensitive Mutation
Brief Title: Icotinib Combined With SBRT for Patients With Metastatic Non-squamous NSCLC With EGFR Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Juan LI, MD, attending physician, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK2017001
Record Dates: First submitted 2017-05-07; First posted 2017-05-15 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer Stage IV
Keywords: EGFR mutation icotinib SBRT
MeSH Terms: conditions — Lung Neoplasms | interventions — icotinib; Radiosurgery

STUDY DESIGN:
Intervention Model Description: icotinib and SBRT treat the lung cancer with egfr mutation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- icotinib+SBRT (Experimental): icotinib 125 milligram,three times a day for 28 days oral administration,12weeks later given the SBRT treatment depended on the outcome of icotinib
  Interventions: Drug: Icotinib; Radiation: SBRT

INTERVENTIONS:
Drug: Icotinib — icotinib 125 milligram three times a day
  Other Names: Icotinib Hydric
Radiation: SBRT — given radiation for the primary lesion
  Other Names: Stereotactic Body Radiation Therapy

SUMMARY:
Many patients with oncogene-driven non-small-cell lung cancer (NSCLC) treated with tyrosine kinase inhibitors experience limited sites of disease progression. For multiple metastases in patients with advanced NSCLC, increased local treatment may benefit to prolong patient survival. This study investigated the benefits of icotinib limited systemic disease progression and continuation of Stereotactic Body Radiation Therapy,in patients with metastatic EGFR-mutant NSCLC.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer morbidity and mortality worldwide. The majority of lung cancer is nonsquamous NSCLC. EGFR tyrosine kinase inhibitors (EGFR-TKI) is a effective first-line treatment for EGFR mutations non-squamous NSCLC treatment.Icotinib is the first EGFR-TKI,and have been proved efficiently in the treatment of lung cancer, and SBRT become a main therapy for the primary lesion,Accordingly, we have come to a scientific hypothesis that icotinib combination with SBRT might be a better treatment strategy for stageIV non-squamous NSCLC patients with EGFR mutation. It can improve the PFS of stage ⅢB/Ⅳ non-squamous NSCLC patients with EGFR mutation . The primary endpoint is disease-free time to progression (PFS). The secondary study endpoint is objective response rate (ORR), disease control rate (DCR),overall survival(OS) safety and quality of life (QOL). Through this study lay the foundation for further exploration of the non-squamous NSCLC first-line treatment in patients with EGFR mutation strategy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of primary lung carcinoma, non-squamous histology with EGFR mutation.
* Stage disease according to the 7th Edition of the American Joint Committee on Cancer staging system
* Not received radiotherapy, chemotherapy or other biological treatment
* Measureable disease
* Life expectancy of>=12 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Absolute neutrophil count (ANC)>=2,500/mm^3
* Hemoglobin>=9.0 g/dL
* Total bilirubin<=1.5 x upper limit of normal(ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate transaminase [AST]) and serum glutamic pyruvic transaminase (SGPT) (alanine transferase [ALT])<=2.5 x ULN in patients without liver or bone metastases; <5 x ULN in patients with liver or bone metastases
* Cockcroft-Gault calculated creatinine clearance of>=45 ml/min or creatinine<=1.5 x ULN
* Prothrombin time (PT)<=1.5 x ULN
* Partial thromboplastin time (PTT)<=ULN
* Negative pregnancy test done<=7 days prior to randomization, for women of childbearing potential only
* Provide informed written consent
* Willing to return to Sichuan cancer hospital for follow-up
* Willing to provide tissue and blood samples for correlative research purposes

Exclusion Criteria:

* Mixed, non-small cell and small cell tumors or mixed adenosquamous carcinomas with a predominant squamous component
* Known allergic to EGFR TKI any ingredients
* Prior chemotherapy or treatment for metastatic non-small cell lung cancer
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive, per MD discretion
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy<=3 years prior to randomization;
* Ongoing or active infection, symptomatic congestive heart failure , cardiac arrhythmia, psychiatric illness/social situations, or any other medical condition that would limit compliance with study requirements
* History of bleeding diathesis or coagulopathy
* Inadequately controlled hypertension (systolic blood pressure of>150 mmHg or diastolic pressure>100 mmHg on anti-hypertensive medications)
* Serious non-healing wound, ulcer, bone fracture, or have undergone a major surgical procedure, open biopsy, or significant traumatic injury <=28 days or core biopsy <=7 days prior to randomization
* Pregnancy or breast-feeding women
* Other situation which researchers think that doesn't fit into the group

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-02 (Estimated); Primary Completion 2017-11-02 (Estimated); Study Completion 2019-05-02 (Estimated)

PRIMARY OUTCOMES:
progression free survival | four weeks
  the time to disease to progression according the RESCIT

SECONDARY OUTCOMES:
object responsible rate | four weeks
  the proportion the patients have receives the complete remission and partial remission

CONTACTS AND LOCATIONS:
Overall Officials: juan li, MD, Principal Investigator — Sichuan Cancer Hospital and Research Institute

IPD SHARING:
Plan to Share IPD: No